CLINICAL TRIAL: NCT00385164
Title: The Utility of 18-Fluorodeoxyglucose Positron Emission Tomography (FDG-PET) for Radiation Treatment Planning in Non-Small Cell Lung Cancer (NSCLC)
Brief Title: The Utility of FDG-PET for Radiation Treatment in NSCLC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: Calgary Health Region (Other)
Responsible Party: Sponsor
Other Study IDs: 20328; E-20328
Record Dates: First submitted 2006-10-04; First posted 2006-10-06 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2011-08

CONDITIONS: Lung Neoplasms; Positron Emission Tomography
Keywords: lung neoplasms; positron emissions tomography; radiotherapy planning
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

INTERVENTIONS:
Procedure: PET/CT scan for RT planning

SUMMARY:
Patients planned for radical radiation for NSCLC will undergo conventional CT stimulation and also PET/CT scans for definition of radiation target volumes

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer to receive radical radiation

Exclusion Criteria:

* unable to tolerate PET/CT scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-small cell lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Harold P Lau, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (1):
- Tom Baker Cancer Centre, Calgary, Alberta, Canada